# Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

Clinical Trials.gov Identifier: NCT04156399

# **Principal Investigator:**

Judith Schlaeger, PhD, CNM, LAc, FAAN

University of Illinois at Chicago, College of Nursing Department of Women, Children and Family Health Science

#### Co-Investigators:

Ardith Doorenbos, PhD, RN, University of Illinois at Chicago College of Nursing,
Department of Biobehavioral Health Science

Crystal Patil, PhD, University of Illinois at Chicago College of Nursing, Department of Women, Children and Family Health Science

Alana Steffen, PhD, University of Illinois at Chicago College of Nursing, Department of Health Systems Science

Robert Molokie, MD, University of Illinois at Chicago College of Medicine and College of Pharmacy

Hongjin Li, PhD, University of Illinois at Chicago College of Nursing, Department of Biobehavioral Health Science

#### Study Location(s):

University of Illinois at Chicago College of Nursing

845 S. Damen Avenue

Chicago, IL 60612

Version: #2.0

**Date:** 11/12/19

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

Version #2.0 11/12/2019

# **TABLE OF CONTENTS**

| | | | Page |
|--------------|---------|--------------------------------------|------|
| Table | e of Co | ontents | 2 |
| List o | of Abb | reviations | 3 |
| 1.0 | Proied | ct Summary/Abstract | 4 |
| 2.0 | | ground/Scientific Rationale | |
| 3.0 | | ctives/Aims | |
| 4.0 | - | oility | |
| 4.0 | | clusion Criteria | |
| | 4.2 Ex | xclusion Criteria | 7 |
| 5.0 | Subie | ect Enrollment | 7 |
| 6.0 | | / Design and Procedures | |
| 7.0 | | cted Risks/Benefits | |
| 8.0 | • | Collection and Management Procedures | |
| 9.0 | | Analysis | |
| | | • | |
| | | ty Control and Quality Assurance | |
| | | and Safety Monitoring | |
| | | stical Considerations | |
| 13.0 | | latory Requirements | |
| | 13.1 | Informed Consent | 9 |
| | 13.2 | Subject Confidentiality | 9 |
| | 13.3 | Unanticipated Problems | 9 |
| 1 <b>4</b> 0 | | ences | |
| | | S | |
| 1.1. | _ | | |

#### LIST OF ABBREVIATIONS

CON College of Nursing

DMC Data Monitoring Committee

DSMB Data and Safety Monitoring Board
DSMP Data and Safety Monitoring Plan
ICD Informed Consent Document
IRB Institutional Review Board

LAR Legally Authorized Representative
OHRP Office of Human Research Protections

OPRS Office for the Protection of Research Subjects

PI Principal Investigator
SAE Serious Adverse Event
SCD Sickle Cell Disease

SOP Standard Operating Procedure UIH University of Illinois Health

## 1.0 Project Summary/Abstract

Our long-term goal is to demonstrate the effectiveness of acupuncture for the treatment of adults with chronic pain of sickle cell disease (SCD), a debilitating pain syndrome characterized by acute and chronic pain. The objective of this study is to explore the feasibility and acceptability of acupuncture with adult sickle cell patients. We will conduct the study with adults with chronic pain from SCD, 18 years old or greater. They will all receive acupuncture. Treatments will be twice weekly for 5 weeks for 30 minutes. At baseline and post-treatment, subjects will complete measures that include pain, fatigue, anxiety, depressive symptoms, injustice experience, pain catastrophizing, and be interviewed about their feelings about receiving acupuncture. Subjects will also complete a measure of study acceptability, the Protocol Acceptability Scale for Treating SCD with Acupuncture at post-treatment. We will describe the procedures and potential challenges to implementing the acupuncture protocol and the range in the subjects' Acceptability Scale scores. We expect to identify and rectify any procedural problems subjects will report regarding the 10-session study protocol.

Version #2.0 11/12/2019

### 2.0 Background/Scientific Rationale

Every 30 minutes, every day, a person dies from a prescription opioid overdose in the United States (US). Further, opioid use is associated with a myriad of adverse outcomes. Sickle cell disease (SCD) affects millions of people worldwide and is the most common lethal genetic blood disorder in the US, affecting about 100,000 people, mostly people of African and Hispanic background. Pain is the most common complication of SCD and is also a marker of clinical severity. People with SCD are a population living with a high burden of chronic pain, high prescription opioid use, and health care disparities. Many with SCD are treated long term with oral opioids and when hospitalized for acute pain are treated with parenteral opioids.

Given this level of opioid use, it is crucial to consider complementary and integrative health (CIH) therapies as a method to decrease exposure to opioids while maintaining adequate pain control. One CIH therapy shown to be acceptable to people with SCD is acupuncture. Acupuncture typically involves inserting small needles into specific points on the body. It is shown to decrease pain and provide an alternative to opioid use. High propagation of the body of the shown to decrease pain and provide an alternative to opioid use. If successful, our project will drastically improve clinic-based pain management and help to reduce reliance on opioids and prevent opioid use disorder.

#### **Acupuncture**

There are few studies of acupuncture for the treatment of SCD. Two were pediatric studies<sup>5</sup> <sup>6</sup> and both reported pain reduction. A third study, which was an uncontrolled retrospective review, treated a total of 24 inpatient and outpatient adults during acute vaso-occlusive crisis with individualized acupuncture point prescriptions.<sup>7</sup> Nine inpatients received a median of 3 treatments and had a reduction in pain of 2.1 on a 0-10 pain rating scale. Fifteen outpatients received a median of 4 treatments and had up to a 75% reduction in pain. The fourth uncontrolled study treated 10 adults with a total of 16 acute vaso-occlusive crises; subjects reported a decrease in pain in 15 of 16 acute vaso-occlusive crises.<sup>8</sup> Because there have been only two trials on using acupuncture for adults with SCD, it is important to generate data on feasibility, acceptability, and protocol revisions for a future fully powered RCT of a standardized acupuncture protocol.

#### 3.0 Objectives/Aims

**Aim:** To determine the feasibility (recruitment, retention, completion) and acceptability of performing acupuncture on 15 adult subjects with SCD.

**Hypothesis:** Acupuncture therapy will be feasible (80% recruitment, retention, completion) and acceptable to adults with SCD.

**Impact:** Acupuncture therapy has the potential to significantly reduce the pain and associated symptoms of SCD by offering therapy that is complimentary to optimal medical management. Symptom management is critical for reducing disability and improving quality of life for people with SCD.

#### 4.0 Eligibility

Adults with SCD who have had a moderate to severe level of pain (<u>></u>3 on 0-10 scale) related to SCD within the last 3 months, receiving care at the UI Health SCD clinic will be eligible to participate.

#### 4.1 Inclusion Criteria

Adults with SCD who have had a moderate to severe level of pain (<u>></u>3 on 0-10 scale) related to SCD within the last 3 months, receiving care at the UI Health SCD clinic will be eligible to participate.

#### 4.2 Exclusion Criteria

- Pregnancy
- Physically or cognitively unable to complete the study procedures

# 5.0 Subject Enrollment

- The primary providers at the UI Health SCD clinic will determine if a patient is eligible for the study.
- Eligibility will be assessed using the Eligibility Checklist. (See Appendix A for Eligibility Checklist).
- The PI or other key research personnel will give out a flyer describing the study to each eligible patient during clinic visits, and explain the general aspects of the study. The flyer also has a contact number for potential subjects to use if interested.
- Patients who express an interest in the study will meet with the PI or other key research personnel, who will explain the study in detail, answer questions, and obtain informed consent.
- Upon consent, patients will be administered baseline study measures.

#### 6.0 Study Design and Procedures

- This study is an unblinded, uncontrolled feasibility study.
- All subjects will receive acupuncture.
- Baseline measures will be taken prior to insertion of the acupuncture needles.
- The research assistant will confirm the subject's assigned code number before the start of each acupuncture session.
- The subject will lay face up on the acupuncture exam table.
- The acupuncturist will swab each of 18 acupuncture points with alcohol.
- Needle insertion will then be performed with a tapping in technique. The
  needles will be retained for 30 minutes; they will be twirled 3 times throughout
  the treatment. The needles will then be pulled.
- After the 10<sup>th</sup> acupuncture treatment the subject will complete data collection tools.

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

#### 7.0 Expected Risks/Benefits

- Expected Risks: There is a risk of bruising or bleeding after the acupuncture needle is withdrawn. There is a risk that they may experience a negative reaction from acupuncture and thereby experience worse symptoms from participation in the study. If potential subjects are afraid of needles, they may not want to participate although the needles are very small. There is risk that some of the questions in the questionnaires may make the subject uncomfortable, nervous or tired. There is also the risk of loss of privacy or confidentiality, but we will avoid this and all other risks as much as possible.
- Expected Benefits: There may be no benefit to individual subjects, but the knowledge gained from this study is expected to help providers better manage SCD pain by having a better understanding of whether or not acupuncture reduces the pain of SCD.

#### 8.0 Data Collection and Management Procedures

- All data will be collected on paper. All subjects will be assigned a code number and their data will be identified only with that code number. The link of the code numbers to the subject identifiers will be kept separate.
- Data management and preliminary data analysis procedures will be supervised by the contact PI (JS).
- The following measures will be completed by the subjects:

| Table: Acupuncture for Adu | Its with Sickle Cell Disease Questionnaires | | | |
|---|---|---|---|---|
| Construct | Operational Measure | 1 | 2 | Source* |
| Demographic data | Age, sex, race, employment status, comorbidities, marital status, number of household members, annual income, and educational attainment | х | | S |
| PROMIS <sup>13</sup> | Perceptions of pain intensity, global health, <sup>14</sup> pain interference, depressive symptoms, <sup>15</sup> anxiety, <sup>9,10</sup> anger, <sup>15</sup> sleep disturbance, <sup>17</sup> fatigue, <sup>18</sup> and selfefficacy <sup>18,19</sup> over the last 7 days, excellent validity across clinical contexts and high internal consistency across diverse racial-ethnic groups (Cronbach's $\alpha$ = 0.92 – 0.96) <sup>20-23</sup> | X | X | Ø |
| McGill Pain Questionnaire (MPQ) | It also documents pain quality via 78 descriptors, and pain pattern via 9 descriptors. <sup>24</sup> The MPQ has demonstrated good reliability (α=.80). <sup>25</sup> | х | Х | S |
| Pain catastrophizing <sup>24</sup> | 13-item scale; measures dimensions of the cognitive appraisal process of pain catastrophizing (magnification, rumination, helplessness); asked to indicate how much they experienced each item (thought/feeling). <sup>25,26</sup> | х | Х | S |
| Injustice Experiences<br>Questionnaire (IEQ-chr) <sup>27</sup> | 12-items; <sup>11</sup> frequency rating for experiencing particular thoughts and feelings, such as "It all seems so unfair," and "Nothing will ever make up for all that I have gone through." <sup>28-32</sup> | х | | S |
| Credibility/Expectancy<br>Questionnaire <sup>12</sup> | 6-items, feelings about acupuncture treatment expectancy and rationale credibility, test–retest 0.62-0.78, Cronbach's α 0.84-0.85. 12 | Х | | S |
| Protocol Acceptability Scale<br>for Treating SCD with<br>Acupuncture | Assesses the <b>acceptability</b> of all study measures being completed and the study itself being completed. This scale will be measured after the last acupuncture session. <sup>33</sup> | | Х | S |
| Cognitive interview | 9 question interview regarding subject's feelings about receiving acupuncture | Х | Х | I |
| | Source: S = Self-report survey, I= Interview | | | |

Version #2.0  11/12/2019

## 9.0 Data Analysis

 Descriptive statistics will be conducted. Descriptive statistics (frequency, percentage, means, and standard deviations) were summarized at baseline. We reported pain intensity, pain interference and other pain related outcomes before and after the acupuncture intervention.

#### 10.0 Quality Control and Quality Assurance

The study is low risk; therefore, we do not anticipate any serious adverse
events from the acupuncture intervention. The PI will provide oversight for the
de-identification of the data. The PI will review all data collection forms on an
ongoing basis for: data completeness, data accuracy and protocol
compliance.

#### 11.0 Data and Safety Monitoring

- The study is low risk. However, the research team will monitor the safety of subjects during study procedures. In the event of injury related to this research, treatment will be available through the UIC Medical Center. However, the patient or third party payer, if any, will be responsible for payment of this treatment. Patient subjects will remain under the care of their usual provider, who will be available to give them usual care if needed. Any unanticipated problems related to the study procedure will be immediately reported to the IRB.
- Data Security: Each participant will be assigned a code number and their data will be identified only with that code number. Only the PI will have access to the code/master key. All questionnaires will be collected on paper and stored in a locked cabinet in the locked PI's office.

#### 12.0 Statistical Considerations

 This is a feasibility study and has not been powered. The data will be descriptive in nature.

# 13.0 Regulatory Requirements

#### 13.1 Informed Consent

- Informed consent will be obtained either by the PI or other key research
  personnel who have obtained IRB and HIPAA certifications. The RA will
  have been trained by the PI on the informed consent procedures. It will be
  obtained on paper.
- The consent process will be completed in person and in a private area at either the UIH SCD Clinic or the acupuncture exam rooms on the 2<sup>nd</sup> floor CON.

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

- Subjects will be informed that they will receive 2 acupuncture treatments for 30 minutes each week for 5 weeks, for a total of 10 treatments.
- Informed consent documents will be stored in a locked file cabinet in the locked PI's office. The study team will have access to the informed consent documents.

#### 13.2 Subject Confidentiality

- All measures will be completed in a private exam room with soundproof walls on the 2<sup>nd</sup> floor of the UIC CON.
- The link between the research data and code number will be destroyed after all manuscripts are published.

#### 13.3 Unanticipated Problems

 Any unanticipated problems related to the study procedure will be immediately reported to the IRB.

#### 14.0 References

- 1. Seth P, Rudd RA, Noonan RK, Haegerich TM. Quantifying the Epidemic of Prescription Opioid Overdose Deaths. *Am J Public Health*. 2018;108(4):500-502.
- 2. Smith WR, Penberthy LT, Bovbjerg VE, et al. Daily assessment of pain in adults with sickle cell disease. *Ann Intern Med.* 2008;148(2):94-101.
- 3. Smith WR, McClish DK, Dahman BA, et al. Daily home opioid use in adults with sickle cell disease: The PiSCES project. *J Opioid Manag.* 2015;11(3):243-253.
- 4. Mathur VA, Kiley KB, Haywood C, Jr., et al. Multiple Levels of Suffering: Discrimination in Health-Care Settings is Associated With Enhanced Laboratory Pain Sensitivity in Sickle Cell Disease. *The Clinical journal of pain.* 2016;32(12):1076-1085.
- 5. Eshkevari L, Heath J. Use of acupuncture for chronic pain: optimizing clinical practice. *Holist Nurs Pract.* 2005;19(5):217-221.
- 6. Zgierska AE, Burzinski CA, Cox J, et al. Mindfulness Meditation and Cognitive Behavioral Therapy Intervention Reduces Pain Severity and Sensitivity in Opioid-Treated Chronic Low Back Pain: Pilot Findings from a Randomized Controlled Trial. *Pain Med.* 2016;17(10):1865-1881.
- 7. Vickers AJ, Vertosick EA, Lewith G, et al. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. *J Pain.* 2018;19(5):455-474.
- 8. Zeidan F, Vago DR. Mindfulness meditation-based pain relief: a mechanistic account. *Ann N Y Acad Sci.* 2016;1373(1):114-127.
- 9. Bhushan D, Conner K, Ellen JM, Sibinga EM. Adjuvant acupuncture for youth with sickle cell pain: a proof of concept study. *Med Acupunct*. 2015;27(6):461-466.
- Tsai S-L, McDaniel D, Taromina K, Lee MT. Acupuncture for Sickle Cell Pain Management in a Pediatric Emergency Department, Hematology Clinic, and Inpatient Unit. *Med Acupunct*. 2015;27(6):510-514.

Version #2.0 

- 11. Lu K, Cheng MJ, Ge X, et al. A retrospective review of acupuncture use for the treatment of pain in sickle cell disease patients: descriptive analysis from a single institution. *Clin J Pain*. 2014;30(9):825.
- 12. Co LL, Schmitz TH, Havdala H, Reyes A, Westerman MP. Acupuncture: an evaluation in the painful crises of sickle cell anaemia. *Pain.* 1979;7(2):181-185.
- 13. Cook KF, Jensen SE, Schalet BD, et al. PROMIS measures of pain, fatigue, negative affect, physical function, and social function demonstrated clinical validity across a range of chronic conditions. *Journal of clinical epidemiology*. 2016;73:89-102.
- 14. Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. *Qual Life Res.* 2009;18(7):873-880.
- 15. Pilkonis PA, Choi SW, Reise SP, et al. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. *Assessment*. 2011;18(3):263-283.
- 16. Kroenke K, Yu Z, Wu J, Kean J, Monahan PO. Operating characteristics of PROMIS four-item depression and anxiety scales in primary care patients with chronic pain. *Pain Med.* 2014;15(11):1892-1901.
- 17. Yu L, Buysse DJ, Germain A, et al. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. *Behav Sleep Med.* 2011;10(1):6-24.
- 18. Cella D, Riley W, Stone A, et al. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. *J Clin Epidemiol*. 2010:63(11):1179-1194.
- 19. Gruber-Baldini AL, Velozo C, Romero S, Shulman LM. Validation of the PROMIS((R)) measures of self-efficacy for managing chronic conditions. *Qual Life Res.* 2017;26(7):1915-1924.
- 20. Jensen RE, Potosky AL, Reeve BB, et al. Validation of the PROMIS physical function measures in a diverse US population-based cohort of cancer patients. Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. 2015;24(10):2333-2344.
- 21. Deyo RA, Dworkin SF, Amtmann D, et al. Focus article report of the NIH task force on research standards for chronic low back pain. *The Clinical journal of pain.* 2014;30(8):701-712.
- 22. Amtmann D, Cook KF, Jensen MP, et al. Development of a PROMIS item bank to measure pain interference. *Pain*. 2010;150(1):173-182.
- 24. Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. *Pain*. 1975;1(3):277-299.
- 25. Wilkie DJ, Savedra MC, Holzemer WL, Tesler MD, Paul SM. Use of the McGill Pain Questionnaire to measure pain: a meta-analysis. *Nurs Res.* 1990;39(1):36-41.
- 23. Fishbain DA, Gao J, Lewis JE, Zhang L. At Completion of a Multidisciplinary Treatment Program, Are Psychophysical Variables Associated with a VAS

Version #2.0 

- Improvement of 30% or More, a Minimal Clinically Important Difference, or an Absolute VAS Score Improvement of 1.5 cm or More? *Pain Med.* 2016:17(4):781-789.
- 26. Sullivan MJL, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. *Psychol Assessment*. 1995;7(4):524-532.
- 27. Keefe FJ, Lipkus I, Lefebvre JC, et al. The social context of gastrointestinal cancer pain: a preliminary study examining the relation of patient pain catastrophizing to patient perceptions of social support and caregiver stress and negative responses. *Pain.* 2003;103(1-2):151-156.
- 28. Badr H, Shen MJ. Pain catastrophizing, pain intensity, and dyadic adjustment influence patient and partner depression in metastatic breast cancer. *Clin J Pain*. 2014;30(11):923-933.
- 29. Sullivan MJ, Adams H, Horan S, Maher D, Boland D, Gross R. The role of perceived injustice in the experience of chronic pain and disability: scale development and validation. *J Occup Rehabil.* 2008;18(3):249-261.
- 30. Yakobov E, Scott W, Stanish W, Dunbar M, Richardson G, Sullivan M. The role of perceived injustice in the prediction of pain and function after total knee arthroplasty. *Pain.* 2014;155(10):2040-2046.
- 31. Sullivan MJ, Scott W, Trost Z. Perceived injustice: a risk factor for problematic pain outcomes. *Clin J Pain*. 2012;28(6):484-488.
- 32. McParland JL, Eccleston C. "It's Not Fair" Social Justice Appraisals in the Context of Chronic Pain. *Curr Dir Psychol Sci.* 2013;22(6):484-489.
- 33. Sullivan MJ, Davidson N, Garfinkel B, Siriapaipant N, Scott W. Perceived injustice is associated with heightened pain behavior and disability in individuals with whiplash injuries. *Psychological Injury and Law.* 2009;2(3-4):238-247.
- 34. Sullivan MJ, Thibault P, Simmonds MJ, Milioto M, Cantin A-P, Velly AM. Pain, perceived injustice and the persistence of post-traumatic stress symptoms during the course of rehabilitation for whiplash injuries. *Pain.* 2009;145(3):325-331.
- 35. Wilkie DJ, Judge MKM, Berry DL, Dell J, Zong S, Gilespie R. Usability of a computerized PAINReportIt in the general public with pain and people with cancer pain. *J Pain Symptom Manag.* 2003;25(3):213–24.

\_\_\_\_\_

Version #2.0  11/12/2019

#### **APPENDICES**

#### **APPENDIX A:**

# Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study Eligibility Checklist

Yes No

#### Inclusion criteria:

- ≥18 years-old with a diagnosis of SCD
- Had a moderate to severe level of pain (≥3 on 0-10 scale) related to SCD within the last 3 months
- Speaks/reads English
- Receiving care at the UI Health SCD clinic

#### Exclusion criteria:

- Pregnant
- Physically or cognitively unable to complete the study procedures

# **APPENDIX B, MEASURES:**

# **Demographic Measures**

#### Sickle Cell Disease Participant Characteristics

| Variable | Category |
|---------------------|-----------------------------------|
| How old are you | |
| What is your | Single |
| marital status | Married/Partnered |
| | White |
| Mbat is your rass | Black/African-American |
| What is your race | Native American/Alaska Native |
| | Hispanic |
| 10/14: | <40k |
| What is your income | 40-50k |
| income | 50k+ |
| How much | < HS, HS, Vocational School |
| education have | Some college or Associates degree |
| you had? | Bachelor's degree or higher |

 $PROMIS\ Item\ Bank\ v.\,1.0-Pain\ Intensity-Scale$ 

#### Pain Intensity - Scale

Please respond to each item by marking one box per row.

| | In the past 7 days | Had no<br>pain | Mild | Moderate | Severe | Very<br>severe |
|---|---|---|---|---|---|---|
| PAINQU6 | How intense was your pain at its worst? | 1 | 2 | 3 | 4 | 5 |
| PAINQUE | How intense was your average pain? | □<br>1 | 2 | 3 | 4 | 5 |
| | | No pain | Mild | Moderate | Severe | Very<br>severe |
| PAINQU21 | What is your level of pain right now? | 1 | 2 | 3 | 4 | 5 |

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

Version #2.0 11/12/2019

#### Global Health

#### Please respond to each question or statement by marking one box per row.

| | | Excellent | Very<br>good | Good | Fair | Poor |
|---|---|---|---|---|---|---|
| Global01 | In general, would you say your health is: | 5 | 4 | 3 | 2 | 1 |
| Global02 | In general, would you say your quality of life is: | 5 | 4 | 3 | 2 | 1 |
| Global03 | In general, how would you rate your physical health? | 5 | 4 | 3 | 2 | I<br>I |
| Global04 | In general, how would you rate your mental health, including your mood and your ability to think? | 5 | 4 | 3 | 2 | I<br>1 |
| Global05 | In general, how would you rate your satisfaction with your social activities and relationships? | 5 | 4 | 3 | 2 | 1 |
| Grobal09r | In general, please rate how well you carry out your usual social activities and roles. (This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc.) | 5 | 4 | 3 | 2 | 1 |
| | _ | Completely | Mostly | Moderately | A little | Not at all |
| Globalód | To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair? | 5 | 4 | 3 | 2 | 1 |

13 April 2018 © 2010-2018 PROMIS Health Organization (PHO)

Page 1 of 2

#### $\mathsf{PROMIS}^{\circledR} \ \mathsf{Scale} \ v1.2 - \mathsf{Global} \ \mathsf{Health}$

#### In the past 7 days...

| | | | _ | Neve | r | Rarely | Some | times | Ofte | n | Always |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Globalför | How often have you been bothered emotional problems such as feeling depressed or irritable? | g anxiou | | 5 | | 4 | -<br>[ | ] | 2 | | 1 |
| | | | _ | None | e | Mild | Mod | erate | Seve | re | Very<br>severe |
| Clobal08r | How would you rate your fatigue of average? | | | 5 | | 4 | -<br>[ | ] | 2 | | 1 |
| Global07r | How would you rate your pain on average? 0 No pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>pain<br>imaginable |

#### Pain Interference

Please respond to each item by marking one box per row.

In the past 7 days...

| | | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| PAININ1 | How difficult was it for you to take in new information because of pain? | 1 | 2 | 3 | 4 | 5 |
| PAININS | How much did pain interfere with your enjoyment of life? | | 2 | 3 | 4 | 5 |
| PAININS | How much did pain interfere with your ability to participate in leisure activities? | I | 2 | 3 | 4 | 5 |
| PAININ6 | How much did pain interfere with your close personal relationships? | 1 | 2 | 3 | 4 | 5 |
| PAINING | How much did pain interfere with your ability to concentrate? | 1 | 2 | 3 | 4 | 5 |
| PAININ9 | How much did pain interfere with your day to day activities? | 1 | 2 | 3 | 4 | 5 |
| PAININ10 | How much did pain interfere with your enjoyment of recreational activities? | I I | 2 | 3 | 4 | 5 |

 $\hbox{$\mathbb{O}$2008-2013 PROMIS$ Health Organization and PROMIS$ Cooperative Group $$ Page 1$ of 5 $$$ 

| | T | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| PAININ11 | How often did you feel emotionally tense because of your pain? | 1 | 2 | 3 | 4 | 5 |
| PAININ12 | How much did pain interfere with the things you usually do for fun? | 1 | 2 | 3 | 4 | 5 |
| PAININ13 | How much did pain interfere with your family life? | 1 | 2 | 3 | 4 | 5 |
| PAININ17 | How much did pain interfere with your relationships with other people? | 1 | 2 | 3 | 4 | 5 |
| PAININ18 | How much did pain interfere with your ability to work (include work at home)? | 1 | 2 | 3 | 4 | 5. |
| PAININ19 | How much did pain make it difficult to fall asleep? | 1 | 2 | 3 | 4 | 5. |
| PAININ20 | How much did pain feel like a burden to you? | 1 | 2 | 3 | 4 | 5, |
| PAININ22 | How much did pain interfere with work around the home? | 1 | | 3 | 4 | 5 |

©2008-2013 PROMIS Health Organization and PROMIS Cooperative Group 

| | | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| PAININ31 | How much did pain interfere with your ability to participate in social activities? | 1 | | 3 | 4 | 5 |
| PAINING4 | How much did pain interfere with your household chores? | 1 | 2 | 3 | 4 | 5 |
| PAININGS | How much did pain interfere with your ability to make trips from home that kept you gone for more than 2 hours? | <u> </u> | 2 | 3 | 4 | 5 |
| PAININ38 | How much did pain interfere with your enjoyment of social activities? | 1 | 2 | 3 | <u>П</u> | 5. |
| PAININ48 | How much did pain interfere with your ability to do household chores? | 1 | | 3 | 4 | 5 |
| PAININ49 | How much did pain interfere with your ability to remember things? | 1 | | 3 | 4 | 5. |
| PAININ56 | How irritable did you feel because of pain? | | | 3 | 4 | 5. |
| PAININ14 | How much did pain interfere with doing your tasks away from home (e.g., getting groceries, running errands)? | 1 | | 3 | <b>□</b> <sub>4</sub> | 5 |

 $\hbox{$\mathbb{O}$2008-2013 PROMIS$ Health Organization and PROMIS$ Cooperative Group $$  $$$ 

| | In the past 7 days | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| PAININ16 | How often did pain make you feel depressed? | 1 | 2 | 3 | 4 | 5 |
| PAININ24 | How often was pain distressing to you? | 1 | 2 | 3 | 4 | 5 |
| PAININ26 | How often did pain keep you from socializing with others? | 1 | 2 | 3 | 4 | 5 |
| PAININ29 | How often was your pain so severe you could think of nothing else? | 1 | 2 | 3 | 4 | 5 |
| PAININ32 | How often did pain make you feel discouraged? | | 2 | 3 | 4 | 5 |
| PAININ37 | How often did pain make you feel anxious? | | 2 | 3 | 4 | 5 |
| Palnins8 | How often did you avoid social activities because it might make you hurt more? | | 2 | 3 | 4 | 5, |
| PAININ40 | How often did pain prevent you from walking more than 1 mile? | 1 | 2 | 3 | 4 | 5 |
| PAININ42 | How often did pain prevent you from standing for more than one hour? | <u> </u> | 2 | 3 | 4 | 5; |

 $\hbox{$\mathbb{O}$2008-2013 PROMIS Health Organization and PROMIS Cooperative Group} \quad \hbox{}$ 

#### In the past $7~\mathrm{days}...$

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| PAININ46 | How often did pain make it difficult for you to plan social activities? | i | | 3 | 4 | 5 |
| PAININ47 | How often did pain prevent you from standing for more than 30 minutes? | ī | | 3 | 4 | 5 |
| PAININ50 | How often did pain prevent you from sitting for more than 30 minutes? | i<br>i | | 3 | 4 | 5 |
| PAININ61 | How often did pain prevent you from sitting for more than 10 minutes? | I<br>I | | 3 | 4 | 5 |
| PAININS2 | How often was it hard to plan social activities because you didn't know if you would be in pain? | 1 | | 3 | 4 | 5 |
| PAININ53 | How often did pain restrict your social life to your home? | 1 | 2 | 3 | 4 | 5 |
| PAININ55 | How often did pain prevent you from sitting for more than one hour? | i | | 3 | 4 | 5 |
| | In the past 7 days | Never | Once a<br>week or<br>less | Once every<br>few days | Once a day | Every few<br>hours |
| PAININ54 | How often did pain keep you from getting into a standing position? | 1 | 2 | 3 | 4 | 5 |

©2008-2013 PROMIS Health Organization and PROMIS Cooperative Group 

#### LEVEL 2—Depression—Adult\*

\*PROMIS Emotional Distress—Depression—Short Form

| Name: | Age: | Sex: ☐ Male ☐ Female | Date: |
|---|---|---|---|
| If the measure is being completed by an informant, | what is your relation | onship with the individual receiving | g care? |
| In a typical week, approximately how much time do | o you spend with th | ne individual receiving care? | hours/week |
| <u>Instructions:</u> On the DSM-5 Level 1 cross-cutting q<br>weeks you (the individual receiving care) have been<br>down, depressed, or hopeless" at a mild or greater<br>detail and especially how often you (the individual<br>7 days. Please respond to each item by marking ( | n bothered by "no i<br>level of severity. The<br>receiving care) hav | nterest or pleasure in doing things'<br>he questions below ask about these<br>e been bothered by a list of sympto | " and/or "feeling<br>e feelings in more |

| | | | | | | | Clinician<br>Use |
|---|---|---|---|---|---|---|---|
| In the past SEVEN (7) DAYS | | | | | | | |
| | | Never | Rarely | Sometimes | Often | Always | Score |
| 1. | I felt worthless. | <b>1</b> | <b>2</b> | □3 | <b>4</b> | <b>□</b> 5 | |
| | | , | | • | | | |
| 2. | I felt that I had nothing to look forward to. | □ 1 | <b>2</b> | □3 | <b>4</b> | □ 5 | |
| 3. | I felt helpless. | □ 1 | <b>□</b> 2 | □3 | <b>4</b> | □ 5 | |
| 4. | I felt sad. | □ 1 | <b>2</b> | □3 | <b>4</b> | <b>□</b> 5 | |
| 5. | I felt like a failure. | □ 1 | <b>□</b> 2 | □3 | <b>4</b> | □ 5 | |
| 6. | I felt depressed. | □ 1 | <b>1</b> 2 | □3 | <b>4</b> | □ 5 | |
| 7. | I felt unhappy. | □ 1 | <b>2</b> | □3 | <b>4</b> | □ 5 | |
| 8. | I felt hopeless. | □ 1 | <b>2</b> | □3 | <b>4</b> | □ 5 | |
| | | | | | Total/Parti | al Raw Score: | |
| Prorated Total Raw Score: | | | | | | | |
| T-Score: | | | | | | | |

©2008-2012 PROMIS Health Organization (PHO) and PROMIS Cooperative Group.
This material can be reproduced without permission by clinicians for use with their patients.
Any other use, including electronic use, requires written permission of the PHO.

#### Emotional Distress - Anxiety - Calibrated Items

Please respond to each item by marking one box per row.

#### In the past 7 days...

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| EDANX01 | I felt fearful | 1 | 2 | 3 | 4 | 5 |
| EDANX02 | I felt frightened | I<br>I | 2 | 3 | 4 | 5 |
| EDANX03 | It scared me when I felt nervous | 1 | 2 | 3 | 4 | 5 |
| EDANX05 | I felt anxious | 1 | 2 | 3 | 4 | 5 |
| EDANX07 | I felt like I needed help for my anxiety | 1 | 2 | 3 | 4 | 5 |
| EDANX08 | I was concerned about my mental health | 1 | 2 | 3 | 4 | 5 |
| EDANX12 | I felt upset | 1 | 2 | 3 | 4 | 5 |
| EDANX13 | I had a racing or pounding heart | 1 | 2 | 3 | 4 | 5 |
| EDANX18 | I was anxious if my normal routine was disturbed | 1 | | 3. | 4 | 5. |

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| EDANX18 | I had sudden feelings of panic | 1 | 2 | 3 | 4 | 5:- |
| EDANX20 | I was easily startled | 1 | 2 | 3 | 4 | 5 |
| EDANX21 | I had trouble paying attention | 1 | 2 | 3 | 4 | 5 |
| EDANX24 | I avoided public places or activities | 1 | 2 | 3 | 4 | 5 |
| EDANX26 | I felt fidgety | 1 | 2 | 3 | 4 | 5 |
| EDANX27 | I felt something awful would happen | 1 | 2 | 3 | 4 | 5 |
| EDANX30 | I felt worried | 1 | 2 | 3 | 4 | 5 |
| EDANXIII | I felt terrified | 1 | 2 | 3 | 4 | 5 |
| EDANX37 | I worried about other people's reactions to me | 1 | 2 | 3 | 4 | 5 |
| EDANX40 | I found it hard to focus on anything other than my anxiety | 1 | 2 | 3. | 4 | 5, |

27 April 2016  $$^{\circ}$$  2008-2016 PROMIS Health Organization and PROMIS Cooperative Group  $$^{\circ}$$  Page 2 of 3

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| EDANX41 | My worries overwhelmed me | 1 | 2 | 3 | 4 | 5 |
| EDANX44 | I had twitching or trembling muscles | 1 | 2 | 3 | 4 | 5 |
| EDANX46 | I felt nervous | 1 | 2 | 3 | 4 | 5 |
| EDANX47 | I felt indecisive | 1 | 2 | 3 | 4 | 5 |
| EDANX48 | Many situations made me worry | 1 | 2 | 3 | 4 | 5 |
| EDANX49 | I had difficulty sleeping | □<br>1 | 2 | 3 | 4 | 5 |
| EDANX51 | I had trouble relaxing | 1 | 2 | 3 | 4 | 5 |
| EDANX53 | I felt uneasy | 1 | 2 | 3 | 4 | 5 |
| EDANX54 | I felt tense | | 2 | 3 | 4 | 5 |
| EDANX55 | I had difficulty calming down | <u> </u> | 2 | 3 | 4 | 5 |

27 April 2016  $\ensuremath{\mathbb{C}}$  2008-2016 PROMIS Health Organization and PROMIS Cooperative Group — Page 3 of 3

#### Emotional Distress - Anger - Short Form 5a

Please respond to each item by marking one box per row.

#### In the past 7 days...

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| EDANG03 | I was irritated more than people knew | 1 | 2 | 3 | 4 | 5 |
| EDANG09 | I felt angry | 1, | 2 | 3 | 4 | .5 |
| EDANG15 | I felt like I was ready to explode | | 2 | 3 | 4 | 5 |
| EDANG30 | I was grouchy | 1 | 2 | 3 | 4 | .5 |
| EDANG35 | I felt annoyed | | 2 | 3 | 4 | 5 |

#### Sleep Disturbance - Calibrated Items

Please respond to each item by marking one box per row.

#### In the past 7 days...

| | in the past / days | | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| Sleep105 | My sleep was restful | 5 | 4 | 3 | | i |
| Sleep108 | My sleep was light | 1 | 2 | 3 | 4 | 5 |
| Sisep107 | My sleep was deep. | 5 | 4 | 3 | | 1 |
| Sleep108 | My sleep was restless. | 1 | 2 | 3 | 4 | 5 |
| Sleep115 | I was satisfied with my sleep | 5 | 4 | 3 | | 1 |
| Sleep116 | My sleep was refreshing | 5 | 4 | 3 | 2 | 1 |
| 6/eep125 | I felt lousy when I woke up | 1 | 2 | 3 | 4 | 5 |
| Sleep20 | I had a problem with my sleep | 1 | 2 | 3 | 4 | 5 |
| Sieep44 | I had difficulty falling asleep | 1 | | 3 | 4 | 5 |
| Sieep65 | I felt physically tense at bedtime | 1 | 2 | 3 | 4 | 5 |

| | • | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| Sieep67 | I worried about not being able to fall asleep. | 1 | 2 | 3 | 4 | 5 |
| Sieep68 | I felt worried at bedtime | 1 | 2 | 3 | 4 | 5 |
| Sleep89 | I had trouble stopping my thoughts at bedtime. | 1 | 2 | 3 | 4 | 5 |
| Sieep70 | I felt sad at bedtime. | 1 | 2 | 3 | 4 | 5 |
| Sleep71 | I had trouble getting into a comfortable position to sleep | 1 | 2 | 3 | 4 | 5 |
| Sleep72 | I tried hard to get to sleep | | 2 | 3 | 4 | 5 |
| Sleep78 | Stress disturbed my sleep | 1 | 2 | 3 | 4 | 5 |
| Sieepilit | I tossed and turned at night | 1 | 2 | 3 | 4 | 5 |
| Sieep93 | I was afraid I would not get back to sleep<br>after waking up. | | 2 | 3 | 4 | 5 |

28 April 2016  $\ensuremath{\mathbb{C}}$  2008-2015 PROMIS Health Organization and PROMIS Cooperative Group  $\ensuremath{\text{Page 2}}$  of 3

| | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| Sleep110 | I got enough sleep | .5 | 4 | 3 | 2 | 1 |
| Sleep#2 | It was easy for me to fall asleep | 5 | 4 | 3 | 2 | 1 |
| Sleep45 | I laid in bed for hours waiting to fall asleep. | ī | 2 | 3 | 4 | 5 |
| Sleep50 | I woke up too early and could not fall back asleep. | ī | 2 | 3 | 4 | 5 |
| Sleep07 | I had trouble staying asleep | 1 | 2 | 3 | 4 | 5 |
| Sleep90 | I had trouble sleeping | 1 | 2 | 3 | 4 | 5 |
| Sleep92 | I woke up and had trouble falling back to sleep. | 1 | 2 | 3 | 4 | 5 |
| | In the past 7 days | Very poor | Poor | Fair | Good | Very good |
| Sleep109 | My sleep quality was | 5 | 4 | 3 | 2 | 1 |

#### Fatigue - Short Form 6a

Please respond to each question or statement by marking one box per row.

#### During the past 7 days...

| × | | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| 1 | I feel fatigued | | | | | |
| 2 | I have trouble starting things because I am tired | | | | | |
| | In the past 7 days | | | | | |
| 3 | How run-down did you feel on average? | | | | | |
| ā | How fatigued were you on average? | | | | | |
| 5 | How much were you bothered by your fatigue on average? | | | | | |
| 6 | To what degree did your fatigue interfere with your physical functioning? | | | | | |

 $PROMIS^{\textbf{\$}} Item \ Bank \ v1.0 - General \ Self \ Efficacy - Short \ Form \ 4a$ 

#### General Self-Efficacy - Short Form 4a

Please respond to each item by marking one box per row.

For the next set of questions, please read each sentence and rate your level of confidence in managing various situations, problems, and events.

| Rate your level of confidence. | | I am not at<br>all<br>confident | I am a<br>little<br>confident | I am<br>somewhat<br>confident | I am quite<br>confident | I am very<br>confident |
|---|---|---|---|---|---|---|
| GSE11_D | I can manage to solve difficult problems if I try hard enough. | 1 | 2 | 3 | 4 | 5 |
| G8E14_0 | I am confident that I could deal efficiently with unexpected events. | 1 | 2 | 3 | 4 | 5 |
| G6E19_C | If I am in trouble, I can think of a solution. | 1 | 2 | 3 | 4 | 5 |
| GSE20_C | I can handle whatever comes my way | 1 | | 3 | 4 | 5 |

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study



# Injustice Experience Questionnaire

Copyright © 2002 Michael JL Sullivan

| | | | | | IEO |
|---|---|---|---|---|---|
| Name: | | | Age: | Gender: | Date: |
| | | open, they can<br>injury has affec | | on our lives. This sca | ale was designed to |
| experien | ce when | you think abou | t your injury. Using the | nt thoughts and feeling<br>e following scale, plea<br>when you think about | se indicate how |
| <b>0</b> – never | | 1 – rarely | 2 – sometimes | 3 – often | 4 – all the time |
| | 1 | Most people | don't understand how | v severe my condition | is. |
| | 2 | My life will | never be the same. | | |
| | 3 | I am sufferi | ng because of someon | e else's negligence. | |
| | 4 | No one shou | ald have to live this wa | ay. | |
| | 5 | I just want t | o have my life back. | | |
| | 6 | I feel that th | is has affected me in a | n permanent way. | |
| | 7 | It all seems | so unfair. | | |
| | 8 | I worry that | my condition is not be | eing taken seriously. | |
| | 9 | Nothing wil | l ever make up for all | that I have gone throu | ıgh. |
| | 10 | I feel as if I | have been robbed of s | omething very precio | us. |
| | 11 | I am trouble | d by fears that I may i | never achieve my drea | ıms. |
| | | I can't belie | ve this has hannened t | o me | |

... Total

Group Number\_\_\_\_ Study Identification Number\_\_\_\_\_

Please answer each item by indicating the number that best describes your response.

1. At this point, how logical does the acupuncture seem to you?

1 2 3 4 5 6 7 8 9 10 not at all somewhat very logical logical logical

2. At this point, how useful do you think the acupuncture will be in reducing your pain?

1 2 3 4 5 6 7 8 9 10 not at all somewhat very useful useful useful

3. How confident would you be in recommending the acupuncture to a friend who experiences similar problems?

1 2 3 4 5 6 7 8 9 10 not at all somewhat very confident confident

4. By the end of the study period, how much improvement in your pain symptoms do you think will occur?

)% 10% 20% 30% 40% 50% 60% 70% 80% 90% 100%

For the last two questions, close your eyes for a few moments, and try to identify what you really feel about the acupuncture and its likely success. Then answer the following questions:

5. At this point, how much do you really fee! that the acupuncture will help you to reduce your pain symptoms?

1 2 3 4 5 6 7 8 9 10 not at all somewhat very much

6. By the end of the study period, how much improvement in your pain symptoms do you really feel will occur?

)% 10% 20% 30% 40% 50% 60% 70% 80% 90% 100%

# $\overline{\Psi}$

# Pain Catastrophization Questionnaire

Copyright © 1995 Michael II, Sullivar

# CS-FN

| | | | | O <b>L</b> / • |
|---|---|---|---|---|
| Client No.: | Age: | Sex: M() F() | Date: | |
| Everyone experiences painful situations at some point in their lives. Such experiences may include headaches, tooth pain, joint or muscle pain. People are often exposed to situations that may cause pain such as illness, injury, dental procedures or surgery. | | | | |
| below are thirter<br>pain. Using the | d in the types of thoughts and<br>en statements describing differe<br>following scale, please indicate<br>ou are experiencing pain. | nt thoughts and feelin | gs that may be | associated with |
| 0 – not at all 1 | - to a slight degree 2 - to a m | noderate degree 3 – to | a great degree | 4 – all the time |
| When I'm in po | in | | | |
| ı | I worry all the time about wh | ether the pain will end | 1. | |
| 2 | I feel I can't go on. | | | |
| 3 | It's terrible and I think it's no | ever going to get any b | etter. | |
| 4 | It's awful and I feel that it ov | verwhelms me. | | |
| 5 | I feel I can't stand it anymore | ð. | | |
| 6 | I become afraid that the pain | will get worse. | | |
| 7 | I keep thinking of other paint | ful events. | | |
| 8 | I anxiously want the pain to | go away. | | |
| 9 | I can't seem to keep it out of | my mind. | | |
| 10 | I keep thinking about how m | uch it hurts. | | |
| 11 | I keep thinking about how ba | dly I want the pain to | stop. | |
| 12 | There's nothing I can do to re | educe the intensity of | the pain. | |
| 13 | I wonder whether something | serious may happen. | | |
| | Total | | | Undated 11/11 |

#### Part 2: What Does Your Pain Feel Like?

Some of the words below describe your **present** pain. Circle **ONLY** those words that describe it. Leave out any category that is not suitable. Use only a single word on eac appropriate category - the one that applies best.

| 1 Flickering Quivering Pulsing Throbbing Beating Pounding | Jumping Flashing Shooting | 3 Pricking Boring Drilling Stabbing Lancinating | 4 Sharp Cutting Lacerating |
|---|---|---|---|
| 5 | 6 | 7 | 8 |
| Pinching | Tugging | Hot | Tingling |
| Pressing | Pulling | Burning | Itchy |
| Gnawing | Wrenching | Scalding | Smarting |
| Cramping | | Searing | Stinging |
| Crushing | | | |
| 9 | 10 | 11 | 12 |
| Dull | Tender | Tiring | Sickening |
| Sore | Taut | Exhausting | Suffocating |
| Hurting | Rasping | | |
| Aching | Splitting | | |
| Heavy | | | |
| 13 | 14 | 15 | 16 |
| Fearful | Punishing | Wretched | Annoying |
| Frightening | Grueling | Blinding | Troublesome |
| Terrifying | Cruel | | Miserable |
| | Vicious | | Intense |
| | Killing | | Unbearable |
| 17 | 18 | 19 | 20 |
| Spreading | Tight | Cool | Nagging |
| Radiating | Numb | Cold | Nauseating |
| Penetrating | Drawing | Freezing | Agonizing |
| Piercing | Squeezing | | Dreadful |
| | Tearing | | Torturing — |

# Part 3: How Does Your Pain Change with Time?

| 1. | Which word or words | would you use to des | cribe the <u>pattern</u> of | your pain? | |
|---|---|---|---|---|---|
| | 1<br>Continuous<br>Steady<br>Constant | 2<br>Rhythmic<br>Periodic<br>Intermittent | 3<br>Brief<br>Momentary<br>Transient | | |
| 2. | What kinds of things I | relieve your pain? | | | |
| 3. | What kinds of things i | ncrease your pain? | | | |
| Pa | rt 4: How Strong Is Y | Your Pain? | | | |
| Pe | ople agree that the follo | | | | |
| | opie agree that the fone | owing o words represe | ent pain of increasi | ng intensity. | They are: |
| N | 0 1 one Mild | 2 Discomforting | 3 | ng intensity. 4 Horrible | They are: 5 Excruciating |
| То | 0 1 | 2<br>Discomforting | 3<br>Distressing | 4<br>Horrible | 5<br>Excruciating |
| To<br>bes | 0 1 one Mild answer each question | Discomforting below, write the number | 3 Distressing ber of the most app | 4<br>Horrible | 5<br>Excruciating |
| To bes | one Mild answer each question side the question. | Discomforting below, write the numbers your pain right now | 3 Distressing ber of the most app | 4<br>Horrible | 5<br>Excruciating |
| To bes | one Mild answer each question side the question. Which word describes | Discomforting below, write the numbers your pain right now sit at its worst? | 3 Distressing ber of the most app | 4<br>Horrible | 5<br>Excruciating |
| To bes | one Mild answer each question side the question. Which word describes Which word describes | Discomforting below, write the number of your pain right now sit at its worst? | 3 Distressing ber of the most app | 4<br>Horrible | 5<br>Excruciating |
| To be: | one Mild answer each question leads the question. Which word describes Which word describes | Discomforting below, write the number syour pain right now sit at its worst? So it when it is least? So the worst toothache | 3 Distressing ber of the most app ? you ever had? | 4<br>Horrible | 5<br>Excruciating |

# Qualitative Interview Guide Regarding Subject's Feelings about Receiving Acupuncture

- 1. What made you decide to join this study on acupuncture?
  - a. Tell me about any past experiences you had with acupuncture
  - b. Do others in your life use acupuncture?
  - c. Not satisfied with your level of pain?
  - d. Heard acupuncture is used to treat pain.
- 2. What were your expectations for getting acupuncture prior to participating in this study?
- 3. Think about your overall acupuncture experience, how would you describe your experience?
  - a. What do you think was happening in your body?
  - b. Did you learn anything from the process of getting acupuncture? What did you learn?
- 4. Describe how acupuncture affected your pain
  - a. Did anything change about how you think about or relate to your pain after going through acupuncture treatments?
- 5. Did anything about getting acupuncture surprise you?
- 6. How is the acupuncture healthcare experience different from other healthcare experiences you have had?
- 7. How did you feel about the acupuncturist?
  - a. Did the acupuncturist treat any medical issues other than pain? What was that like?
- 8. Tell me the reasons you would or would not continue to get acupuncture in the future.
- 9. Is there anything else you would like us to know about how acupuncture affected you and your overall experience?

#### Protocol Acceptability Scale for Treating Sickle Cell Disease with Acupuncture \* (select the most appropriate answer) 1. Was participating in this study too hard? Not hard at all Somewhat hard Too hard 2. Were the study instructions easy to understand? \_Easy to understand Somewhat hard to understand Too hard to understand 3. Were the study questions easy to see? \_ Easy to see Somewhat hard to see \_ Too hard to see 4. Did you feel rushed to complete this study? Not rushed at all Somewhat rushed Too hard to complete 5. Did you enjoy being in this study? Enjoyed participating Somewhat enjoyed participating \_\_ Did not enjoy participating 6. What did you think of getting acupuncture? \_ I liked it I did not like it \_ I didn't like it or not like it 7. Did you think acupuncture was painful? \_ It was not painful \_\_\_\_ It was painful 8. Would you get acupuncture again? \_ I would get it again I would not get it again 9. Do you think this study will be well received by other adults with sickle cell disease? \_ Others will enjoy being in this study Others will somewhat enjoy being in this study Others will not enjoy being in this study 10. Do you think the study was: Too short \_ Too long Right length

- 1. Eshkevari L, Heath J. Use of acupuncture for chronic pain: optimizing clinical practice. *Holist Nurs Pract.* 2005;19(5):217-221.
- 2. Zgierska AE, Burzinski CA, Cox J, et al. Mindfulness Meditation and Cognitive Behavioral Therapy Intervention Reduces Pain Severity and Sensitivity in Opioid-

Acupuncture for Adults with Sickle Cell Disease (SCD): A Feasibility Study

\*Protocol Acceptability Scale adapted from Wilkie et al. 2003 & Wilkie et al. 2001

- Treated Chronic Low Back Pain: Pilot Findings from a Randomized Controlled Trial. *Pain Med.* 2016;17(10):1865-1881.
- 3. Vickers AJ, Vertosick EA, Lewith G, et al. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. *J Pain.* 2018;19(5):455-474.
- 4. Zeidan F, Vago DR. Mindfulness meditation-based pain relief: a mechanistic account. *Ann N Y Acad Sci.* 2016;1373(1):114-127.
- 5. Bhushan D, Conner K, Ellen JM, Sibinga EM. Adjuvant acupuncture for youth with sickle cell pain: a proof of concept study. *Med Acupunct*. 2015;27(6):461-466.
- 6. Tsai S-L, McDaniel D, Taromina K, Lee MT. Acupuncture for Sickle Cell Pain Management in a Pediatric Emergency Department, Hematology Clinic, and Inpatient Unit. *Med Acupunct*. 2015;27(6):510-514.
- 7. Lu K, Cheng MJ, Ge X, et al. A retrospective review of acupuncture use for the treatment of pain in sickle cell disease patients: descriptive analysis from a single institution. *Clin J Pain*. 2014;30(9):825.
- 8. Co LL, Schmitz TH, Havdala H, Reyes A, Westerman MP. Acupuncture: an evaluation in the painful crises of sickle cell anaemia. *Pain.* 1979;7(2):181-185.
- 9. Pilkonis PA, Choi SW, Reise SP, et al. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. *Assessment*. 2011;18(3):263-283.
- 10. Kroenke K, Yu Z, Wu J, Kean J, Monahan PO. Operating characteristics of PROMIS four-item depression and anxiety scales in primary care patients with chronic pain. *Pain Med.* 2014;15(11):1892-1901.
- 11. Sullivan MJ, Adams H, Horan S, Maher D, Boland D, Gross R. The role of perceived injustice in the experience of chronic pain and disability: scale development and validation. *J Occup Rehabil.* 2008;18(3):249-261.
- 12. Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. *Journal of behavior therapy and experimental psychiatry*. 2000;31(2):73-86.

\_\_\_\_\_

Version #2.0  11/12/2019